CLINICAL TRIAL: NCT03537729
Title: A Randomized Controlled Trial of Visual Cues, Signage, and Spaced-Retrieval Education Within Long Term Care Communities to Assist With Wayfinding
Brief Title: Effects of Visual Cues and Education for People Who Live Within Long Term Care Communities to Assist in Wayfinding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Principal Investigator, Rebecca Davis, Professor, Grand Valley State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P17203009
Record Dates: First submitted 2018-05-04; First posted 2018-05-25 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease; Alzheimer Dementia; Age-Related Memory Disorders; Dementia
Keywords: Alzheimer's disease; Age related memory disorders; Environment design; Long term care; Dementia
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): There will be no modifications to décor or signage in the existing care community, and no education on wayfinding. However, subjects will receive the same testing that is provided for the other arms at the designated time periods.
- Salient Cues (Experimental): Special signs and salient cues will be added to the community along the routes being measured for wayfinding. The cues will be comprised of pictures, objects, and signage.
  Interventions: Behavioral: Salient Cues
- Spaced retrieval education (Experimental): This condition will have signage and cues as in Arm 2 added to the care communities. In addition, a spaced retrieval (SR) memory intervention strategy will be implemented individually for each resident participating in the study to help them remember the presence and function of the environmental wayfinding cues.
  Interventions: Behavioral: Salient Cues; Behavioral: Spaced Retrieval Education

INTERVENTIONS:
Behavioral: Salient Cues — Salient cues are those that capture the individual's attention. Information that is complex, novel, and difficult to identify takes more processing resources than those that are simple and familiar. Cues such as pictures and wall hangings, along with bright and meaningful signs, will be placed at key decision points within the senior communities.
  Arms: Salient Cues; Spaced retrieval education
Behavioral: Spaced Retrieval Education — Spaced Retrieval (SR) is an evidence-based memory strategy that is used to teach individuals with memory loss new or previously known information. In this study, participants in Arm 3 will receive twelve 30-minute educational sessions to help them use the salient cues to find their way.
  Arms: Spaced retrieval education

SUMMARY:
The ability to find one's way in the world is known as wayfinding. Many older adults who live in senior communities, such as independent living and assisted living residences, find wayfinding very challenging. Often times, these communities are not designed in a way that helps people find their way very easily. When people cannot find their way, they can get lost, be dependent upon others for getting out and about, or even be afraid to leave their rooms. The purpose of this study is to find out if distinctive signs and decorative elements, along with a special type of education called Spaced-Retrieval education, help residents in these communities find their way more effectively. Twelve senior communities will be assigned by chance to one of three conditions, including: 1) control - no change (the community stays the same); 2) signs and decorative elements enhanced; and 3) signs, decorative elements, and special education added. After agreeing to be in the study, the participants will be asked to find their way to certain places in their community four times over a year. Some people will be asked to participate in educational sessions on wayfinding. In addition, some people will be asked to wear a location tracker, (like a fitness tracker), for four weeks during the year. How well people find their way, along with how much they travel about within the communities, will be compared between the three groups. It is hypothesized that those in the communities with special signs and decorative elements will find their way more effectively than those in the control communities. It is also hypothesized that participants in the communities with the special education intervention will find their way better than those without the education. Finally, it is hypothesized that participants in the communities with signs and cues and education will travel about further distances than those in the control communities. The results of the study can help people who have a tendency to get lost find their way more effectively in their community, and this could result in more independence.

DETAILED DESCRIPTION:
The ability to locate and travel successfully to a destination, known as wayfinding, is a significant problem for older adults with cognitive disorders. Relocating to a new residence such as independent or assisted living is a time in which older adults with cognitive problems are most vulnerable to experiencing wayfinding problems. Often these communities are not designed to facilitate wayfinding as they are complex, confusing, and lack distinctiveness. Wayfinding problems can cause individuals' worlds to shrink, leading to a smaller life space (the spatial extent of travel within the community), decreased engagement, and dependence upon others for activities of daily living. The overall goal of the proposed project is to assess the contribution of salient visual cues and Spaced Retrieval (SR) on wayfinding ability and life space in older adults with wayfinding problems who live in senior communities. Salient cues, such as vivid pictures, statues and bright, distinctive signage can make senior residential communities more memorable and distinctive. This study has three specific aims: a) to examine the effect of salient cues with and without SR on wayfinding ability initially and over time in older adults who have wayfinding deficits in senior communities; and b) To determine the effects of salient visual cues and SR on life space; and c) to determine subject characteristics that are most amenable to the intervention; wand which subject characteristics place persons at risk for less responsiveness to the intervention so that the intervention can be appropriately targeted. There are three arms to the clinical trial to which nine care communities will be randomly assigned, including Arm 1 (control; no change to the care community); Arm 2 (colorful and familiar objects and signage placed within the care community); and Arm 3 (Arm 2 cues plus SR). Participants will be individuals within the communities who exhibit problems finding their way. They will be asked to find their way repeatedly to specific destinations over a period of a year. Wayfinding performance, including how fast the participants find the test location and the errors they make compared between study Arms. Life space will also be measured and compared between Arms. It is hypothesized that individuals who are in care communities which are enhanced with salient cues will improve wayfinding when compared to care communities without salient cues. In addition, Spaced Retrieval, which is an evidence-based memory strategy, is hypothesized to positively influence subjects' use of the cues and improve wayfinding performance. Finally, it is hypothesized that wayfinding ability will correlate with life space. The long term goals of this research are to test an evidence based intervention to enhance senior residences so that older adults who have wayfinding problems can more easily learn and remember their environments so that they can maintain independence.

ELIGIBILITY:
Inclusion Criteria:

* Age 62 or older;
* Wayfinding impairment identified by the subject or staff and exhibited at baseline, including problems finding their way among three defined locations (these may differ among care communities);
* Ability to move self either independently by walking or using mobility aids (self-mobile; any mobility aids are acceptable)
* Ability to communicate with researchers and follow directions
* Ability to see and read signs in English.

Exclusion Criteria:

* Chronic health conditions that impair the ability to participate in the study, such as severe chronic obstructive pulmonary disease (COPD) (limiting movement) or terminal illness;
* Signs of rapid deterioration in health during the past 6 months as evidenced by staff communication or medical records.

Min Age: 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Davis, PhD, Principal Investigator — Grand Valley State University
Locations (2):
- United States (2):
  - Grand Valley State University, Allendale, Michigan
  - Brush Development, Chardon, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from approximately 138 subjects from nine senior living communities. The final dataset will include de-identified data, including certain demographics, wayfinding data, and cognitive tests. We will make the data and associated documentation (code book, description of variables) available to users in Scholarworks. ScholarWorks@GVSU is an open-access repository maintained by the Grand Valley State University (GVSU) Libraries. It is anticipated that the data would be available after the PI has published the final results, or within two years of the completion of the study. The repository will have the de-identified data set, along with a description of each variable and any statistical formulas used to create the variable.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within six months of final publication of the data.
Access Criteria: We will make the data and associated documentation (code book, description of variables) available to users in Scholarworks. ScholarWorks@GVSU is an open-access repository maintained by the GVSU Libraries. It is anticipated that the data would be available after the PI has published the final results, or within two years of the completion of the study. The repository will have the de-identified data set, along with a description of each variable and any statistical formulas used to create the variable.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen senior living communities were enrolled and randomized to one of three arms between June 2019 and June 2022. Residents (individual participants) were recruited from each community. The first participant was enrolled on June 12, 2019 and the last was enrolled on June 16, 2022. There was a significant pause in enrollment due to the COVID-19 pandemic.
Pre-assignment Details: Senior living communities were randomized, with individual participants clustered within senior living communities.
Units Other Than Participants: Senior Living Communities
Period: Overall Study
Arm/Group | Control | Salient Cues | Spaced Retrieval Education
Started | 55; 5 Senior Living Communities | 62; 5 Senior Living Communities | 55; 5 Senior Living Communities
Completed Month 0 | 43; 5 Senior Living Communities | 57; 5 Senior Living Communities | 50; 5 Senior Living Communities
Completed Month 1 | 39; 5 Senior Living Communities | 54; 5 Senior Living Communities | 47; 5 Senior Living Communities
Completed Month 3 | 35; 5 Senior Living Communities | 52; 5 Senior Living Communities | 46; 5 Senior Living Communities
Completed Month 6 | 27; 3 Senior Living Communities | 33; 3 Senior Living Communities | 25; 3 Senior Living Communities
Completed | 25; 3 Senior Living Communities | 28; 3 Senior Living Communities | 21; 3 Senior Living Communities
Not Completed | 30; 2 Senior Living Communities | 34; 2 Senior Living Communities | 34; 2 Senior Living Communities
Not completed — Death | 2 | 2 | 7
Not completed — Withdrawal by Subject | 3 | 3 | 0
Not completed — Subject Moved | 8 | 5 | 4
Not completed — Investigator determined not in best interest for subject to continue | 1 | 0 | 0
Not completed — COVID-19 Site Restrictions | 11 | 15 | 18
Not completed — Decline in Health | 5 | 9 | 4
Not completed — Determined Ineligible | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data were collected only on the participant level.
Units Other Than Participants: Senior Living Communities
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Salient Cues | Spaced Retrieval Education | Total
Number analyzed (Participants) | 43 | 57 | 50 | 150
Number analyzed (Senior Living Communities) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.37 (5.16) | 85.59 (6.00) | 84.26 (6.49) | 85.07 (5.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 46 | 39 | 118
  Male | 10 | 11 | 11 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 56 | 50 | 149
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 43 | 56 | 50 | 149
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 57 | 50 | 150
Adjusted Wayfinding Speed [Mean (Standard Deviation); unit: feet per second] — Subjects walked three pre-specified routes in the senior living community (simple, moderate, and complex). They were timed as they walked the route using a computer application called DOTT. Rest periods, elevator wait times and errors (wrong turns) were indicated in DOTT as the participant traversed the route. The adjusted wayfinding speed was calculated as the length of the route in linear feet divided by time in seconds the subject took to walk the route, minus rest periods and elevator wait times, plus 120 seconds added per error.
  feet per second
    Adjusted Wayfinding Speed (Low complexity route) | 1.58 (1.36) | 2.91 (2.63) | 1.57 (1.05) | 2.08 (1.98)
    Adjusted Wayfinding Speed (moderate complexity route) | 1.33 (1.05) | 1.61 (0.89) | 1.37 (0.74) | 1.45 (0.90)
    Adjusted Wayfinding Speed (high complexity route) | 1.29 (0.88) | 0.95 (0.48) | 1.12 (0.60) | 1.10 (0.67)
Wayfinding accuracy [Mean (Standard Deviation); unit: proportion of possible errors on a route] — Accuracy was measured via proportion of errors, calculated as number of errors made by a participant when walking a pre-specified route divided by number of possible errors on a route. Errors were defined as a subject making a wrong turn at a decision point, or a U-turn in a hallway the wrong direction. Higher value reflects lower accuracy (higher proportion of errors).
  proportion of possible errors on a route
    Wayfinding accuracy (low complexity route) | 0.12 (0.20) | 0.11 (0.25) | 0.08 (0.15) | 0.11 (0.20)
    Wayfinding accuracy (moderate complexity route) | 0.14 (0.15) | 0.10 (0.13) | 0.10 (0.12) | 0.11 (0.13)
    Wayfinding accuracy (high complexity route) | 0.12 (0.12) | 0.21 (0.13) | 0.14 (0.13) | 0.16 (0.13)
Tinetti Life Space [Mean (Standard Deviation); unit: score on a scale] — Tinetti's Nursing Home Life-Space Diameter scale measures life space on the scale from 0 to 100. Higher scores represent larger life space, indicating movement throughout the senior living residence and leaving the building. Low scores indicate less movement within the building (a smaller life-space).
  score on a scale | 47.63 (12.34) | 52.61 (13.34) | 57.96 (16.48) | 53.25 (15.10)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Wayfinding Speed (Feet Per Second)
Description: Subjects walked three pre-specified routes in the senior living community (simple, moderate, and complex). They were timed as they walked the route using a computer application called DOTT. Rest periods, elevator wait times and errors (wrong turns) were indicated in DOTT as the participant traversed the route. The adjusted wayfinding speed was calculated as the length of the route in linear feet divided by time in seconds the subject took to walk the route, minus rest periods and elevator wait times, plus 120 seconds added per error.
Time Frame: Average over months 1, 3, 6, and 12
Population: Participants walking routes
Measure: Least Squares Mean (Standard Error); unit: feet per second
Arm/Group | Control | Salient Cues | Spaced Retrieval Education
Number analyzed (Participants) | 43 | 57 | 50
feet per second
  Adjusted Wayfinding Speed (low complexity route) | 2.32 (0.15) | 2.87 (0.14) | 2.33 (0.14)
  Adjusted Wayfinding Speed (moderate complexity route) | 1.83 (0.09) | 1.97 (0.09) | 1.81 (0.09)
  Adjusted Wayfinding Speed (high complexity route) | 1.42 (0.09) | 1.48 (0.08) | 1.57 (0.08)
Statistical Analysis 1: Comparison: Control vs Salient Cues; The null hypothesis was that means of two arms on the low complexity route are equal, the alternative was that means were not equal; Test type: Superiority — Power was based on planned 12 sites and effect size Cohen's d=0.42 for pairwise differences between arms, intraclass correlation coefficient of 0.0012, and reduction in variance due to adjustment for baseline and repeated measures with correlation of 0.4 between pairs of measures. The sample size requirement was 38 per group, or 114 total for power of .80 in two-sided tests at .05 level of significance; p < .01, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Covariates included baseline value of the outcome, age, sex, and cognition score at baseline, and use of wheelchair on the route; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [0.18 to 0.91], Standard Error of Mean 0.19 — Cues minus control
Statistical Analysis 2: Comparison: Control vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .96, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.35 to 0.37], Standard Error of Mean 0.18 — Spaced retrieval minus control
Statistical Analysis 3: Comparison: Salient Cues vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < .01, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.89 to -0.18], Standard Error of Mean 0.18 — Spaced retrieval minus cues only
Statistical Analysis 4: Comparison: Control vs Salient Cues; The null hypothesis was that means of two arms on the moderate complexity route are equal, the alternative was that means were not equal; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .23, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.09 to 0.38], Standard Error of Mean 0.12 — Cues minus control
Statistical Analysis 5: Comparison: Control vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .90, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.25 to 0.22], Standard Error of Mean 0.12 — Spaced retrieval minus control
Statistical Analysis 6: Comparison: Salient Cues vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .17, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.38 to 0.07], Standard Error of Mean 0.11 — Spaced retrieval minus cues only
Statistical Analysis 7: Comparison: Control vs Salient Cues; The null hypothesis was that means of two arms on the high complexity route are equal, the alternative was that means were not equal; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .58, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.16 to 0.28], Standard Error of Mean 0.11 — Cues minus control
Statistical Analysis 8: Comparison: Control vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 7]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .15, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.06 to 0.37], Standard Error of Mean 0.11 — Spaced retrieval minus control
Statistical Analysis 9: Comparison: Salient Cues vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 7]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .37, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.11 to 0.29], Standard Error of Mean 0.10 — Spaced retrieval minus cues only

2. Primary Outcome: Wayfinding Accuracy on Simple Route
Description: Accuracy was measured via proportion of errors, calculated as number of errors made by a participant when walking a pre-specified route divided by number of possible errors on a route. Errors were defined as a subject making a wrong turn at a decision point, or a U-turn in a hallway the wrong direction. Higher value reflects lower accuracy (higher proportion of errors).
Time Frame: Average over months 1, 3, 6, and 12
Population: Participants who completed wayfinding.
Measure: Least Squares Mean (Standard Error); unit: proportion of errors made on route
Arm/Group | Control | Salient Cues | Spaced Retrieval Education
Number analyzed (Participants) | 43 | 57 | 50
proportion of errors made on route | 0.083 (0.01) | 0.046 (0.01) | 0.053 (0.01)
Statistical Analysis 1: Comparison: Control vs Salient Cues; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .04, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.07 to -0.01], Standard Error of Mean 0.02 — Cues minus control
Statistical Analysis 2: Comparison: Control vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .10, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.07 to 0.01], Standard Error of Mean 0.02 — Spaced retrieval minus control
Statistical Analysis 3: Comparison: Salient Cues vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .69, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.03 to 0.04], Standard Error of Mean 0.02 — Spaced retrieval minus cues only

3. Primary Outcome: Wayfinding Accuracy on Moderate and Complex Routes
Description: as for outcome 2
Time Frame: Average over months 1, 3, 6, and 12
Population: Participants who completed wayfinding assessments.
Measure: Least Squares Mean (Standard Error); unit: proportion of errors made on route
Arm/Group | Control | Salient Cues | Spaced Retrieval Education
Number analyzed (Participants) | 43 | 57 | 50
proportion of errors made on route
  Wayfinding accuracy on moderate route | 0.21 (0.03) | 0.14 (0.02) | 0.12 (0.02)
  Wayfinding accuracy on complex route | 0.10 (0.02) | 0.13 (0.02) | 0.08 (0.02)
Statistical Analysis 1: Comparison: Control vs Salient Cues; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = 0.04, Generalized mixed model analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Ratio of mean proportions of errors = 0.65, 95% CI 2-sided [0.44 to 0.99] — Ratio of mean proportion of errors for cues divided by proportion of errors for control. Log of the mean was estimated from generalized linear mixed effects models for each arm. The difference between logs of means for two arms was exponentiated
Statistical Analysis 2: Comparison: Control vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .01, Generalized mixed model analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Ratio of mean proportions of errors = 0.59, 95% CI 2-sided [0.39 to 0.90] — Ratio of mean proportion of errors for spaced retrieval divided by proportion of errors for control. Log of the mean was estimated from generalized linear mixed effects models for each arm. The difference between logs of means was exponentiated
Statistical Analysis 3: Comparison: Salient Cues vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .61, Generalized mixed model analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Ratio of mean proportions of errors = 0.90, 95% CI 2-sided [0.60 to 1.35] — Ratio of mean proportion of errors for spaced retrieval divided by proportion of errors for cues. Log of the mean was estimated from generalized linear mixed effects models for each arm. The difference between logs of means was exponentiated
Statistical Analysis 4: Comparison: Control vs Salient Cues; [analysis description as in outcome 1, analysis 7]; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .26, Generalized mixed model analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Ratio of mean proportions of errors = 1.26, 95% CI 2-sided [0.84 to 1.88] — Ratio of mean proportion of errors for cues divided by proportion of errors for control. Log of the mean was estimated from generalized linear mixed effects models for each arm. The difference between logs of means was exponentiated
Statistical Analysis 5: Comparison: Control vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 7]; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .25, Generalized mixed model analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Ratio of mean proportions of errors = 0.79, 95% CI 2-sided [0.53 to 1.19] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: Salient Cues vs Spaced Retrieval Education; [analysis description as in outcome 1, analysis 7]; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .03, Generalized mixed model analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Ratio of mean proportions of errors = 0.63, 95% CI 2-sided [0.42 to 0.94] — [estimate comment as in outcome 3, analysis 3]

4. Secondary Outcome: Life Space
Description: Tinetti's Nursing Home Life-Space Diameter scale measures life space on the scale from 0 to 100. Higher scores represent larger life space.
Time Frame: Average over months 1, 3, 6, and 12
Population: Participants who completed life space assessments.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Salient Cues | Spaced Retrieval Education
Number analyzed (Participants) | 43 | 57 | 50
score on a scale | 52.63 (1.36) | 50.91 (1.20) | 51.84 (1.28)
Statistical Analysis 1: Comparison: Control vs Salient Cues; The null hypothesis was that means of two arms are equal, the alternative was that means were not equal; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .31, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Covariates included baseline value of the outcome, age, sex, and cognition score at baseline; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-5.03 to 1.60], Standard Error of Mean 1.69 — Cues minus control
Statistical Analysis 2: Comparison: Control vs Spaced Retrieval Education; The null hypothesis was that means of two arms are equal, the alternative was that means were not equal; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .66, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Covariates included baseline value of the outcome, age, sex, and cognition score at baseline; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-4.23 to 2.66], Standard Error of Mean 1.75 — Spaced retrieval minus control
Statistical Analysis 3: Comparison: Salient Cues vs Spaced Retrieval Education; The null hypothesis was that means of two arms are equal, the alternative was that means were not equal; Test type: Superiority — Sample size was determined by power analysis for the adjusted wayfinding speed; p = .57, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Covariates included baseline value of the outcome, age, sex, and cognition score at baseline; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [-2.30 to 4.17], Standard Error of Mean 1.65 — Spaced retrieval minus cues only

ADVERSE EVENTS:
Time Frame: One year from baseline.
Arm/Group | Control | Salient Cues | Spaced Retrieval Education
All-Cause Mortality (participants affected / at risk) | 7/55 | 2/62 | 9/55
Serious Adverse Events (participants affected / at risk) | 4/55 | 9/62 | 6/55
Other Adverse Events (participants affected / at risk) | 6/55 | 7/62 | 11/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=55) | Salient Cues (N=62) | Spaced Retrieval Education (N=55)
Hospitalization (General disorders) | 4 (4) | 7 (9) | 5 (5) — Participant was hospitalized for unspecified reason.
Fall with injury (General disorders) | 0 (0) | 3 (3) | 2 (2) — A fall was reported with non-specific injury.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=55) | Salient Cues (N=62) | Spaced Retrieval Education (N=55)
Outpatient Hospitalization (General disorders) | 0 (0) | 1 (1) | 1 (1) — Went to emergency department or other outpatient area for unknown reason but was discharged home the same day.
Fall with injury (General disorders) | 2 (2) | 3 (3) | 3 (3) — A fall with resulting injury, non specified.
Fall without injury (General disorders) | 2 (2) | 3 (3) | 2 (2) — A fall was reported but no injury sustained.
Minor Illness (General disorders) | 1 (1) | 0 (0) | 4 (4) — Minor illness was reported but not specified.
Too fatigued (General disorders) | 1 (1) | 0 (0) | 1 (1) — Participant became too fatigued to continue in the study.

LIMITATIONS AND CAVEATS:
The study was conducted during a world-wide pandemic, causing cessation of study activities and participant attrition. The sample was a convenience sample; those who participated may be different than those who did not. We were unable to recruit a diverse sample due to the lack of diversity in the independent living and assisted living settings; this limits generalizability of the findings. The intraclass correlation was higher than expected due to the routes being community specific.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03537729/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03537729/SAP_001.pdf
  • Informed Consent Form (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT03537729/ICF_002.pdf